CLINICAL TRIAL: NCT00714103
Title: A Phase I Study of 8-Chloro-Adenosine in Previously Treated Patients With Chronic Lymphocytic Leukemia /Small Lymphocytic Lymphoma
Brief Title: 8-Chloro-Adenosine in Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0144; NCI-2012-01679 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Leukemia; Chronic Lymphocytic Leukemia
Keywords: Leukemia; Chronic Lymphocytic Leukemia; CLL; 8-Chloro-Adenosine; purine analogues; Cancer
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — 8-chloroadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 8-Chloro-Adenosine (Experimental): Starting dose for first cohort of patients 45 mg/m2 intravenous over 1 hr daily for 5 days every 4 weeks (± 3 days).
  Interventions: Drug: 8-Chloro-Adenosine

INTERVENTIONS:
Drug: 8-Chloro-Adenosine — 45 mg/m^2 intravenous over 1 hour daily for 5 days every 4 weeks (± 3 days).

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of the drug 8-chloro-adenosine that can be given in the treatment of chronic lymphocytic leukemia (CLL). Another goal is to learn how effective the drug is at treating leukemia.

DETAILED DESCRIPTION:
8-Chloro-adenosine is a new drug similar to other drugs already approved by the FDA for the treatment of CLL and other types of cancer. 8-Chloro-adenosine belongs to a class of chemotherapy drugs called purine analogues that work to treat cancer by their ability to interfere with cancer cell metabolism, causing cell death.

If you are eligible, you will receive 8-chloro-adenosine as an infusion into a vein once a day for five days in a row. Each infusion will take about 1 hour. This 5-day treatment will be repeated every 4 weeks (± 3 days) (1 course).

This is a dose escalation study. Patients treated on this study will be treated in groups of 3. The first group will receive the lowest dose of the drug. If the type, number, and severity of any side effects experienced are acceptable, the next group of 3 patients will receive the next higher dose of drug. The dose of drug will be increased for each new group until the highest safe dose is found.

For your first course only, you will have blood tests (about 1 tablespoon) on Day 3 and Day 5 of treatment to monitor for safety. After that, you will have weekly (± 3 days) evaluations and routine blood tests (about 1 tablespoon) in the clinic at University of Texas MD Anderson Cancer Center (UTMDACC). During these evaluations, you will also have a physical exam and be asked about any side effects you may have experienced. You will be evaluated for improvement in your CLL. If your disease is stable or responding to treatment, you may continue with treatment. If your disease improves to the point that your doctor feels that you are in complete remission, he or she will request you to have a bone marrow biopsy to confirm complete remission.

If your disease is worsening and it appears that the treatment is not helping you, then you will stop treatment with 8-chloro-adenosine and may begin other treatment at the direction of your treating doctor. If you have unacceptable side effects, you may be taken off treatment.

If you stop treatment, you will be evaluated in the clinic and have routine blood tests (about 1 tablespoon) once a week for the first month, twice a month for the next 2 months, then once a month from then on. During these evaluations, you will have a physical exam and be asked about any side effects you may have experienced. If you begin other treatment, your scheduled follow-up will end.

This is an investigational study. 8-Chloro-adenosine is not approved by the FDA and is not commercially available. A total of up to 28 patients will take part in this study. All will be enrolled and treated at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of chronic lymphocytic leukemia and must be previously treated with at least one prior treatment regimen, including a purine-analogue based treatment.
2. Patients must be Rai Stage III or IV OR Rai Stage 0-II and have one or more criteria for active disease as defined by the NCI-Working Group as: a) weight loss of more than 10% in the last 6 months; b) fatigue; c) fever or night sweats without evidence of infection; d) progressive anemia or thrombocytopenia; e) progressive lymphocytosis with a lymphocyte doubling time </= 6 months; or f) marked hypogammaglobulinemia or paraproteinemia.
3. All patients must have a Zubrod performance status of </= 2.
4. All patients must be age >/= 18 years.
5. Patients may not receive concurrent treatment for their CLL and must have been off treatment (chemotherapy, immunotherapy, or radiotherapy) for 4 weeks prior to treatment on this study and recovered from toxic effects of that therapy.
6. All patients must have adequate renal function indicated by serum creatinine </=2.5x upper limits of normal (ULN) and adequate liver function indicated by ALT or AST </= 2.5x ULN AND total bilirubin </= 2.5x ULN.
7. All patients must have a pre-treatment platelet count of >/= 50,000 /µl and not require transfusion to maintain this platelet count unless thrombocytopenia is due to marrow infiltrated with disease.
8. All patients or appropriate surrogate must provide informed consent.

Exclusion Criteria:

1. Patients with active uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia purpura.
2. Patients with active uncontrolled fungal, bacterial, or viral infection.
3. Patients who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity and Maximum Tolerated Dose | 4 weeks
  During first course of treatment blood tests on Days 3 and 5; then weekly (± 3 days) evaluations and routine blood tests. Toxicity evaluation completed four weeks following initial 8-Chloro-adenosine administration.

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org